CLINICAL TRIAL: NCT04865965
Title: Effects of a Single Bout of Exercise on Transcriptomics and Metabolomics in Adipose Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000139
Record Dates: First submitted 2021-04-13; First posted 2021-04-29 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Metabolic Complication
Keywords: adipose tissue transcriptomics; adipose tissue metabolomics; peripheral blood mononuclear cell transcriptomics; obesity; exercise
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Bout of Exercise (Experimental): Exercising for 60 minutes at 55-60% of VO₂ peak
  Interventions: Procedure: Acute Bout of Exercise
- No Exercise (No Intervention): No Exercise Session

INTERVENTIONS:
Procedure: Acute Bout of Exercise — Exercising for 60 minutes at 55-60% of VO₂ peak
  Arms: Acute Bout of Exercise

SUMMARY:
The purpose of this study is to determine the effects of a single bout of exercise on changes in the genes and small molecules in blood and fat tissue, before and after a bout of exercise. This research may contribute to a better understanding of the beneficial effects of exercise on the body.

DETAILED DESCRIPTION:
The national and international prevalence of both obesity and type 2 diabetes has risen dramatically over the last few decades, increasing the need for new therapies to treat these conditions. An established treatment for type 2 diabetes and obesity are regular physical activity and exercise. It has been shown that one single session of exercise can lead to adaptations in the blood and in tissues that improve systemic homeostasis overtime; while acute changes in skeletal muscle also play a critical role in these effects, changes in the adipose tissue and in the peripheral mononuclear cells (PBMCs) that may also contribute to this improvement. However, the beneficial effects of exercise on metabolism through these other tissues have not been intensively investigated.

The investigators hypothesize that a single session of exercise will result in changes to white adipose tissue, including changes in metabolites and gene expression, as well as changes in PBMCs, and that these adaptations may play an important role to improve metabolic homeostasis.

This hypothesis stems from the investigator's animal-based studies, which have led to the exciting discoveries that 1) exercise training-induced adaptations to subcutaneous white adipose tissue (scWAT) result in significant improvements in whole-body glucose tolerance and insulin sensitivity (1), and 2) the mechanism for this effect may be due to auto-, para-, or endocrine effects of novel exercise-induced circulating factors coming from adipose tissue. Thus, being able to further understand, and potentially mimick, these exercise-induced changes to scWAT could lead to novel therapies for obesity and type 2 diabetes.

Given the great interest in exercise mimetics as treatments for diabetes and obesity, it is essential to determine if a single session of exercise alters metabolites as well as gene expression in the scWAT in human subjects with obesity. To determine if a single session of exercise leads to changes in PBMCs, PBMC transcriptomics will be analyzed. This analysis will determine how exercise affects the number of specific cell types in the blood that can regulate metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60 years
* Body mass index (BMI) ≥30.0 ± 0.1 and ≤40.0 ± 0.1 kg/m2
* HbA1c ≤ 5.7 ± 0.1%
* No history of diabetes (type 1 and type 2)
* In good general health with no conditions that could influence the outcome of the trial, and in the judgment of the investigator is a good candidate for the study based on review of available medical history, physical examination and clinical laboratory evaluations
* Willing to adhere to the protocol requirements for the duration of the study

Exclusion Criteria:

* Exercises frequently i.e. ≥ 150 minutes per week of moderate intensity or ≥ 75 min high intensity.
* Blood glucose rises ≥140mg/dl at 2 hours after OGTT on Visit 1
* Use of weight loss medications (i.e. GLP-1 agonists)
* Use of any medications related to diabetes
* Use of beta-blockers
* Use of anticoagulation and aspirin
* Use of agents that affect hepatic glucose production such as beta adrenergic agonists, xanthine derivatives
* Currently pregnant or breastfeeding
* Current smoker
* Heart or lung disease
* Acute infection, including COVID-19 (current or recent infection of COVID-19 in the previous 3 months)
* Any hospitalization due to COVID-19.
* Severe hypertension (systolic >160 mmHg or diastolic >90 mmHg)
* Inability to exercise for any reason
* Any known contraindication to exercise testing based on current ACSM guidelines (5)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Transcriptome in white adipose tissue | Baseline; 2 hours
  Gene transcription changes in RNA-based expression within subcutaneous adipose tissue
Metabolome in fat | Baseline; 2 hours
  Changes in concentration of metabolites within subcutaneous adipose tissue

SECONDARY OUTCOMES:
Transcriptomic changes in peripheral blood mononuclear cell in people with obesity | Baseline; 2 hours
  Gene transcription changes in RNA-based expression within peripheral blood mononuclear cells

CONTACTS AND LOCATIONS:
Overall Officials: Roeland JW Middelbeek, MD, Principal Investigator — Joslin Diabetes Center; Laurie Goodyear, PhD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States